CLINICAL TRIAL: NCT01421628
Title: The Effectiveness of a Trainings Program on ADL Performance, Physical Fitness, Wellbeing, and Nocturnal Cramp in Elderly People
Brief Title: Enhancement of Physical Fitness in Older Adults
Acronym: NLC2010
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanze University of Applied Sciences Groningen (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Hank Hallegraeff Msc,PT, PhD student
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HanzeUnlc
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2010-12

CONDITIONS: Pain; Physical Impairment
Keywords: older adults; exercise; stretching; mobility
MeSH Terms: conditions — Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise (Experimental)
  Interventions: Other: Fitness exercise program

INTERVENTIONS:
Other: Fitness exercise program — Exercise program, daily frequency, duration of 6 weeks.

SUMMARY:
Ageing is related to a decrease in physical fitness, disability and age related symptoms like nocturnal leg cramps (NLC). Our research is focused on the enhancement of physical activity and mobility to increase physical fitness and decrease disability and nocturnal cramp in older adults.

DETAILED DESCRIPTION:
The ageing population leads to an increase of chronic disease and disability and to a decrease of physical activity and ADL performance. This circle can be reversed by physical exercise to increase physical fitness.

The goal of this research is to establish the effects of a trainings program on ADL performance, physical fitness and nocturnal cramps. Furthermore the characteristics from participants who benefit from the program will be investigated by the research.

The study design is a randomized intervention study. Participants are elderly people, age 65 years and older, without cognitive impairment.

Intervention: The intervention is a physical trainings program. The intensity is moderate, the frequency is daily and the total duration is 6 weeks. The control group will be provided with an education program.

Main parameters are: physical fitness, nocturnal cramp severity and frequency.

ELIGIBILITY:
Inclusion Criteria:

* For patients to be included in our study, they had to experience regular episodes of NLC and are in good mental health.
* The participants had to agree to the study protocol and complete the program.
* After eligibility was verified, written informed consent was obtained.

Exclusion Criteria:

* Older adults taking quinine or sleep medication and those with orthopedic problems or with severe medical problems and co morbidity, which can cause muscular spasms and/or cramps.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Physical fitness | six weeks
  Strength, balance
ADL performance | six weeks
  Performance based ADL test
Well being | six weeks
  Questionnaires like SF-36
Nocturnal cramps | Six weeks
  Visual analogue scale (VAS)

SECONDARY OUTCOMES:
Frequency nocturnal cramp | Six weeks
  Number of cramp attacks per day.

CONTACTS AND LOCATIONS:
Overall Officials: Hank Hallegraeff, PT, MSc, Principal Investigator
Locations (1):
- Kinese Fysiotherapeuten, Appingedam, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Hallegraeff JM, van der Schans CP, de Ruiter R, de Greef MH. Stretching before sleep reduces the frequency and severity of nocturnal leg cramps in older adults: a randomised trial. J Physiother. 2012;58(1):17-22. doi: 10.1016/S1836-9553(12)70068-1. PMID 22341378